CLINICAL TRIAL: NCT05764551
Title: he Application of DNA Methylation for Patients Who Had Hepatocellular Carcinoma With Normal Serum Alpha-fetoprotein
Brief Title: The Application of Serum DNA Methylation for Patients With HCC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chiayi Christian Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB2022051
Record Dates: First submitted 2023-02-28; First posted 2023-03-10 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-02

CONDITIONS: Hepatocellular Carcinoma
Keywords: DNA methylation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- DNA methylation (Experimental): The enrolled individuals with HCC would receive serum DNA methylation test before their treatment (including all kinds of recommened HCC treatment). Then regularly serum DNA methylation test would be done at 4th~8th weeks, 16th week, 32th week and 48th week. If the enrolled patients did not have HCC recurrence during at 48th week. The regular check of serum DNA methylation would be canceled. The enrolled patients would be observed till 96th week. If there is any recurrence during 48~96th week, one time of serum DNA methylation would be checked at the time of recurrence. The observation and intervention would be completed at 96th week.
  Interventions: Diagnostic Test: Serum DNA methylation

INTERVENTIONS:
Diagnostic Test: Serum DNA methylation — Serum DNA methylation

SUMMARY:
The goal of this single-arm prospective study is to evaluate the application of serum DNA methylation for HCC patients with normal alpha-fetoprotein. The main question it aims to answer is

. Is the dynamic change of serum DNA methylation correlated to recurrence or treatment response of HCC

DETAILED DESCRIPTION:
The enrolled individuals with HCC and normal serum alpha-fetoprotein level would receive serum DNA methylation test before their treatment (including all kinds of recommened HCC treatment). Then regularly serum DNA methylation test would be done at 4th~8th weeks, 16th week, 32th week and 48th week. If the enrolled patients did not have HCC recurrence during at 48th week. The regular check of serum DNA methylation would be canceled. The enrolled patients would be observed till 96th week. If there is any recurrence during 48~96th week, one time of serum DNA methylation would be checked at the time of recurrence. The observation and intervention would be completed at 96th week.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 20 years old
* The diagnosis of hepatocellular carcinoma (HCC) according to AASLD 2018 clinical guidelines or histology report
* Individuals with HCC and normal serum alpha-fetorpotein level (<20 ng/ml)
* Individuals who could sign informed consent

Exclusion Criteria:

* The histology report revealed non-HCC, HCC mixed with cholangiocarcinoma or sarcomatoid HCC
* Individuals with HCC and other concurrent malignancies
* Individuals with chronic kidney disease who could not tolerate contrast-enhanced dynamic images
* Individuals ever receiving any organ transplantation
* Individuals with HIV infection
* Individuals who could not able to understand and sign informed consent

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-03-28 (Estimated); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
The correlation between serum DNA methylation and HCC recurrence or treatment response | 96 weeks
  The correlation between serum DNA methylation and HCC recurrence or treatment response

CONTACTS AND LOCATIONS:
Overall Officials: Po-Yueh Chen, M.D, Principal Investigator — Ditmanson Medical Foundation Chiayi Christian Hospital
Locations (1):
- Ditmanson Medical Foundation Chiayi Christian Hospital, Chiayi City, Taiwan

IPD SHARING:
Plan to Share IPD: No